CLINICAL TRIAL: NCT04861909
Title: Long-term Efficacy, Visual Performance and Patient Reported Outcomes With a Trifocal Intraocular Lens: Six-year Follow-up
Brief Title: Long-term With a Trifocal Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Qvision, Ophthalmology Department (Other)
Collaborators: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: QVI-20-02
Record Dates: First submitted 2021-02-19; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Cataract
Keywords: Multifocal intraocular lens; Long-term; Safety; Efficacy; Defocus curve; Light distortion
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AT LISA tri 839MP: Patients implanted with AT LISA tri 839MP
  Interventions: Device: AT LISA tri 839MP

INTERVENTIONS:
Device: AT LISA tri 839MP — Non interventional study

SUMMARY:
The main aims of this study were to evaluate the patient reported outcomes (PROs), safety and efficacy, after 6-year (66 - 78 months) from the binocular implantation of the AT LISA tri 839MP. A secondary aim was to evaluate new metrics such as contrast sensitivity defocus curves and light distortion analysis.

DETAILED DESCRIPTION:
Retrospective cross-sectional study with two stages:

• Phone call interview:

First stage included patient reported outcomes of visual function, spectacle independence and satisfaction through questionnaires conducted by a phone call in all the patients implanted in our center with AT LISA 839MP from March 2014 to June 2015 (n=92) which accomplished inclusion / exclusion criteria and were able to be contacted by phone (n=62).

The incidence of Nd-YAG capsulotomy was retrospectively evaluated through the revision of the medical history, in patients for which capsulotomy was conducted in our center, or a question, for those treated in another center.

• Study visit:

Second stage included the consecutive invitation of these phone interviewed patients to a visit in our center for a long-term visual performance assessment up to accomplish the required sample size (n=37).

Corrected and uncorrected monocular visual acuities were the primary end-points for testing non-inferiority hypothesis in comparison to 12-month follow-up mean results reported in the literature. Secondary variables of assessment were contrast sensitivity defocus curve and light distortion analysis.

ELIGIBILITY:
Inclusion Criteria:

* Phone call interview:

  * Patients of either sex, 45 years of age or older at the time of surgery and less than 80 years of age at the time of the phone call.
  * Patients implanted bilaterally with the AT LISA 839MP MIOL in the capsular bag.
  * No surgical complications reported in the clinical history that could affect postoperative visual acuity: damage to the capsular bag, intraocular hemorrhage, etc.
  * Operated between 66 months from the first implanted eye and up to 78 months from the surgery of the second eye
  * Patient able to hear, understand and give express consent orally.
* Study visit:

  * To have participated in the first stage of the study corresponding to the phone call interview.
  * Irregular astigmatism in either eye measured with corneal tomography (total high-order corneal aberrations at 4 mm < 0.5 μm).
  * Patient able to read, understand and provide a written informed consent form.
  * Sufficient availability, willingness, skills, and cognitive awareness to comply with follow-up/study procedures and study visits.

Exclusion Criteria:

* Phone call interview:

  * Any eye disease documented in the patient's clinical history that may potentially cause a loss of visual acuity or diplopia: Active or recurrent pathology of the anterior segment (chronic uveitis, iritis, iridocyclitis, rubeosis iridis, uncontrolled glaucoma, etc.), retinal or optic nerve pathologies such as diabetic retinopathy, macular degeneration, etc.
  * Eye surgery (including laser refractive surgery) performed before or after the operation with the intraocular lens.
* Study Visit:

  * PCO ≥ 2 according to surgeon criteria that produces a loss of CDVA ≥ 0.2 logMAR
  * Any eye disorder that can potentially cause a loss of visual acuity or diplopia: Active or recurrent pathology of the anterior segment (chronic uveitis, iritis, iridocyclitis, rubeosis iridis, uncontrolled glaucoma, etc.), retinal or optic nerve pathologies such as diabetic retinopathy, macular degeneration, etc.
  * Eye surgery (including laser refractive surgery) performed before or after the operation with the intraocular lens.
  * Use of systemic or ocular medications that may affect vision in the last 6 months.
  * Subjects who participate in any clinical trial or research with drugs or medical devices within 30 days prior to entry into this research and/or during the period of participation in this research.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients implanted with AT Lisa Tri from March 2014 to June 2015
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Monocular visual acuity | 6 years
  Visual acuity measured with and without best corrected distance subjective refraction in logMAR scale, lower value meaning better results.

SECONDARY OUTCOMES:
Contrast sensitivity defocus curve in logCS | 6 years
  Contrast Sensitivity measured at different vergence distances with Multifocal Lens Analyzer (www.defocuscurve.com) in logCS scale, higher value meaning better results.
Light distortion analysis in percentage | 6 years
  Light Distortion Analyzer (CEORLab, University of Minho, Braga, Portugal) in Percentage, higher percentage meaning poorer results.
Visual Function Questionnaire (VF-14) | 6 years
  Patient reported outcomes evaluation of difficulties related to visual function in daily life activities (Scale ranging from 0 - 100, higher values meaning better results)
Patient-Reported Spectacle Independence Questionnaire (PRSIQ) | 6 years
  Patient reported outcomes of spectacle independence showing descriptive results of percentage of patients using need of glasses, often wear and comfortably without wear
Satisfaction, Photic Phenomena and Operated again | 6 years
  Independent questions not associated with a validated questionnaire showing descriptive results of percentage of patients satisfied with their vision, the bothersome to photic phenomena and the likely to be operated again.

CONTACTS AND LOCATIONS:
Locations (1):
- Qvision, Vithas Virgen del Mar Hospital, Almería, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04861909/Prot_SAP_000.pdf